CLINICAL TRIAL: NCT00000944
Title: A Phase I Trial of the Safety, Tolerance, and Pharmacokinetics of Oral Indinavir Co-Administered With Lamivudine (3TC) and Zidovudine (ZDV) in HIV-1-Infected Pregnant Women During Gestation and Post Partum, and in Their Infants Post Maternal Dosing
Brief Title: A Study to Evaluate the Safety and Tolerance of Combination Anti-HIV Drug Therapy (Indinavir, Lamivudine, and Zidovudine) in HIV-Positive Pregnant Women and Their Infants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Purpose: Prevention
Other Study IDs: ACTG 358; PACTG 358; 10606 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections; Pregnancy
Keywords: Pregnancy; Pregnancy Complications, Infectious; Drug Therapy, Combination; Zidovudine; HIV Protease Inhibitors; Lamivudine; Indinavir; Disease Transmission, Vertical; Anti-HIV Agents
MeSH Terms: conditions — HIV Infections; Pregnancy Complications, Infectious | interventions — Indinavir; Lamivudine; Zidovudine

INTERVENTIONS:
Drug: Indinavir sulfate
Drug: Lamivudine
Drug: Zidovudine

SUMMARY:
The purpose of this study is to determine if a combination anti-HIV drug treatment regimen of indinavir plus lamivudine (3TC) plus zidovudine (ZDV) is effective in treating HIV and in reducing the chances of passing HIV from mother to child. This study will also examine if this combination is well tolerated by HIV-positive pregnant women and if a combination of 3TC plus ZDV is safe for newborns.

Previous studies in adults and children have shown that indinavir plus 3TC plus ZDV can reduce the amount of HIV in the blood. Most HIV-positive pregnant women usually take ZDV to treat HIV and to reduce the chances of giving HIV to their babies. The combination of drugs in this study may be more effective than ZDV alone.

DETAILED DESCRIPTION:
Despite the dramatic reduction of perinatal HIV transmission following the administration of ZDV to mothers and infants, new, more effective strategies are needed. An increasing number of women may require combination antiretroviral therapy for their own disease because they may be resistant to ZDV, may have high viral loads, or may have previously transmitted HIV to an infant while on ZDV monotherapy. The initiation of triple combination therapy, including a protease inhibitor indinavir, during gestation may be the most effective in reducing maternal virus load prior to delivery, thereby potentially benefitting both mother and child.

Women:

Antepartum (until active labor): Indinavir plus 3TC plus ZDV. Intrapartum (active labor until cord clamping): 3TC plus ZDV. Postpartum (after cord clamped to 12 weeks): Indinavir plus 3TC plus ZDV.

Infants:

3TC plus ZDV as soon as oral intake is tolerated (preferably within 12 hours of birth) and continuing for 6 weeks.

[AS PER AMENDMENT 1/27/99: For maternal dosing, one Combivir tablet bid can be substituted for the individual formulation of 3TC and ZDV. For mothers who receive Combivir during the antepartum period, Combivir is held during labor and delivery, and the separate formulations of ZDV and 3TC are used. Patients who prematurely discontinue study treatment should continue to be followed on study for the duration of the study.]

ELIGIBILITY:
Inclusion Criteria

Women may be eligible for this study if they:

* Are HIV-positive.
* Have been pregnant for 14-28 weeks (are in your 1st or 2nd trimester).
* Have a normal ultrasound exam when they are screened for the study.
* Are able to drink 6 glasses of water a day throughout the study.
* Are at least 13 years old (need consent of parent or guardian if under 18).

Exclusion Criteria

Women will not be eligible for this study if they:

* Cannot take 3TC or ZDV.
* Have an active opportunistic (HIV-associated) or bacterial infection at study entry.
* Have chronic diarrhea.
* Have epilepsy or cancer.
* Are pregnant with more than 2 children (triplets, etc.)
* Have risk factors for premature birth, or other problems with their pregnancy.
* Have any immediate life-threatening illness.
* Have severe anemia or other illness for which they require blood products.
* Have a history of chronic liver or kidney disease.
* Plan to breast-feed.

Min Age: 13 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24
Dates: Study Completion 2003-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diana Wara, Study Chair; Yvonne Bryson, Study Chair; Ruth Tuomala, Study Chair
Locations (4):
- United States (4):
  - UCSF Pediatric AIDS CRS, San Francisco, California
  - HMS - Children's Hosp. Boston, Div. of Infectious Diseases, Boston, Massachusetts
  - Jacobi Med. Ctr., The Bronx, New York
  - Montefiore Med. Ctr. - AECOM, The Bronx, New York